CLINICAL TRIAL: NCT05059912
Title: Humanized CD7 CAR T-cell Therapy for R/R CD7+ T Cell Lymphoma
Brief Title: CD7 CAR T-cell for R/R CD7+ T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Affiliated Hospital of Jiangnan University (Other); Affiliated Zhongshan Hospital of Dalian University (Other); The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD7T
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Refractory and Relapsed T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 positive relapsed or refractory T cell lymphoma (Experimental): Humanized CD7 CAR-T cells intravenously infused to patient with R/R T-NHL[ at a dose of (0.5- 5)x10^6 CD7 CAR-T cells/kg
  Interventions: Biological: Humanized CD7 CAR-T cells

INTERVENTIONS:
Biological: Humanized CD7 CAR-T cells — Patients will receive infusion of CAR T-cells targeting CD7 to confirm the safety and efficacy of CD7 CAR T-Cells in CD7+ relapsed or refractory T cell lymphoma

SUMMARY:
This is a prospective, open-label, multiple center and single arm phase 2 study to evaluate the efficacy and safety of T cells expressing humanized CD7 chimeric antigen receptors treatment for patients with refractory/relapsed CD7 positive T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. R/R T-NHL with measurable (≧1.5cm) lesions confirmed by pathological immunohistochemistry or flow cytometry
3. The expressions of both CD4 and CD8 are negative in patients with bone marrow involved
4. The Eastern Cooperative Oncoloy Group (ECOG) physical condition score ≤ 2 points
5. The main organ functions need to meet the following conditions:

   A.Left ventricular ejection fraction ≥50% B.Creatinine ≤132umol/l or creatinine clearance ≥60 ml/min C.ALT and AST≤2.5 upper limitation of normal D.T-BIL≤2.0mg/dl E.SpO2 > 90%
6. Results of pregnant test should be negative, and agree to conception control during treatment and 1 year after CAR-T infusion
7. Expected survival exceeds 3 months
8. Written informed consent could be acquired

Exclusion Criteria:

1. Immunosuppressant medications or steroids were used within 2 weeks before cell collection, or need to use steroids or immunosuppressant medications more than two years
2. Patients with uncontrolled active infection
3. Active hepatitis B or hepatitis C infection
4. Patients with HIV infection
5. Severe acute or chronic graft-versus-host disease (GVHD)
6. Participated in any other drug research clinical trials within 30 days before enrollment
7. Prior CAR-T cells therapy within 3 months before enrollment
8. Prior allogeneic hematopoietic stem cell transplantation within 6 months before enrollment
9. Uncontrolled other tumor
10. Women in pregnancy, lactation or planning to become pregnant
11. The researcher considers inappropriate to participate in this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-08-03 (Estimated); Study Completion 2024-08-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 1 year
  Number of patients who achieved response (complete response and partial response ) after treatment of CD7 CAR-T cell. Response will be assessed using the Lugano criteria.
Number of Adverse Events | 1 year
  Adverse events are evaluated with CTCAE V5.0

SECONDARY OUTCOMES:
Complete relapse rate(CR) | 1 year
  Number of patients who achieved complete response after treatment by CD7 CAR-T cell.
Duration of overall response (DOR) | 1 year
  Duration of overall response will be assessed from the CAR-T cell infusion to progression, death or last follow-up.
Progression-free survival(PFS) | 1 year
  PFS will be assessed from the CAR-T cell infusion to progression, death or last follow-up.
Overall survival(OS) | 1 year
  OS will be assessed from the CAR-T cell infusion to death or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D&Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No